CLINICAL TRIAL: NCT02495025
Title: Developing and Testing a New Model for Telephone-based Early Childhood Developmental Screening and Care Coordination in Vulnerable Populations
Brief Title: Testing the Effectiveness of Telephone-based Early Childhood Developmental Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Paul Chung, Associate Professor of Pediatrics, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-000509
Record Dates: First submitted 2015-07-08; First posted 2015-07-13 (Estimated); Results first posted 2019-10-14 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-09

CONDITIONS: Child Development; Developmental Disabilities; Ambulatory Care; Screening
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: Participants were randomized individually at the time of enrollment, to receive either telephone-based developmental screening and care coordination, through 2-1-1 Los Angeles, in addition to usual care, or usual care alone. Primary outcomes were measured at 6 months after enrollment.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telephone-based screening (Experimental): Families randomized to the intervention arm will be connected with 211 Los Angeles for completion of developmental screening over the phone. Screening will consist of three structured, validated, parent-report tools: the Parental Evaluation of Developmental Status (PEDS), the PEDS Developmental Milestones (PEDS:DM), and the Modified Checklist for Autism in Toddlers (M-CHAT). If any developmental or behavioral concerns are present, the care coordinator at 211 Los Angeles will make appropriate referrals for developmental evaluation and intervention services. A copy of the care plan generated from 211 will be sent to the child's primary care provider and included in the medical record.
  Interventions: Behavioral: Telephone-based developmental screening and care coordination
- Usual care (No Intervention): Children randomized to the control group will report for their well-child care visits as scheduled, and will receive clinic-based developmental screening and care coordination. Any developmental or behavioral concerns will be directed to the child's pediatrician, as is the current clinical recommendation.

INTERVENTIONS:
Behavioral: Telephone-based developmental screening and care coordination
  Arms: Telephone-based screening

SUMMARY:
The purpose of this research study is to test the effectiveness of telephone-based early childhood developmental screening and care coordination, compared to usual care in a primary care pediatrics clinic. Investigators randomized 152 participants to one of two study arms, with the intervention families receiving developmental screening over the phone, and control families receiving usual care with their pediatricians.

DETAILED DESCRIPTION:
Although the American Academy of Pediatrics (AAP) recommends universal early childhood developmental screening as part of routine well-child care, there have been many studies documenting that many pediatricians do not follow the AAP guidelines. One intervention that has the potential to improve care, especially for low-income families, is centralized, telephone-based developmental screening, and care coordination for families whose children have developmental or behavioral concerns. 2-1-1 Los Angeles developed such an intervention and this study aims to test its effectiveness, in partnership with a local community clinic, using a randomized, controlled study design. Investigators partnered with the Clinica Oscar A Romero, a federally-qualified health center in Los Angeles, serving predominantly low-income Latino families. Investigators hope to enroll up to 300 families in the study. Eligible families will have children ages 12 to 42 months of age who receive well-child care at the clinic. As investigators obtain informed consent and enroll families, they will randomize study participants into intervention and control groups. Intervention group families will be transferred to 211 Los Angeles to complete developmental screening over the phone, while control group families will go to their pediatricians for well-child care as usual.

ELIGIBILITY:
Inclusion Criteria:

* child receives well-child care at the clinic
* child is not already receiving intervention services for a developmental disability
* parent speaks Spanish or English well enough to be interviewed

Exclusion Criteria:

* child is younger than 12 months or older than 42 months at time of enrollment
* child is already receiving intervention services for a developmental disability
* parent is unable to speak Spanish or English well enough to be interviewed

Ages: 12 Months to 42 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 152 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Chung, MD, MS, Principal Investigator — Universilty of California, Los Angeles
Locations (1):
- Clinica Oscar A Romero, Los Angeles, California, United States

REFERENCES:
- [Derived] Nelson BB, Thompson LR, Herrera P, Biely C, Arriola Zarate D, Aceves I, Estrada I, Chan V, Orantes C, Chung PJ. Telephone-Based Developmental Screening and Care Coordination Through 2-1-1: A Randomized Trial. Pediatrics. 2019 Apr;143(4):e20181064. doi: 10.1542/peds.2018-1064. PMID 30894408

RESULTS

PARTICIPANT FLOW:
Groups:
- Telephone-based Screening: Families randomized to the intervention arm will be connected with 211 Los Angeles for completion of developmental screening over the phone. Screening will consist of three structured, validated, parent-report tools: the Parental Evaluation of Developmental Status (PEDS), the PEDS Developmental Milestones (PEDS:DM), and the Modified Checklist for Autism in Toddlers (M-CHAT). If any developmental or behavioral concerns are present, the care coordinator at 211 Los Angeles will make appropriate referrals for developmental evaluation and intervention services. A copy of the care plan generated from 211 will be sent to the child's primary care provider and included in the medical record.
  Telephone-based developmental screening and care coordination
Period: Overall Study
Arm/Group | Telephone-based Screening | Usual Care
Started | 77 | 75
Completed | 51 | 61
Not Completed | 26 | 14
Not completed — Lost to Follow-up | 21 | 14
Not completed — Withdrawal by Subject | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telephone-based Screening | Usual Care | Total
Number analyzed (Participants) | 77 | 75 | 152
Age, Continuous [Mean (Standard Deviation); unit: months] | 25.7 (9.5) | 23.3 (7.9) | 24.5 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 43 | 76
  Male | 44 | 32 | 76
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Latino or Hispanic | 72 | 71 | 143
  Race/ethnicity: White, non-Hispanic | 1 | 0 | 1
  Race/ethnicity: Black of African-American | 3 | 0 | 3
  Race/ethnicity: Other | 0 | 1 | 1
  Race/ethnicity: Unknown | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Screened With a Validated Tool
Description: We will measure whether developmental screening was done using a validated instrument, as recommended by the AAP. Specific screening instruments include the Parental Evaluation of Developmental Status (PEDS), the PEDS: Developmental Milestones (PEDS:DM), the Ages and Stages Questionnaires (ASQ), and/or the Modified Checklist for Autism in Toddlers (MCHAT), Revised version.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Telephone-based Screening | Usual Care
Number analyzed (Participants) | 77 | 75
Participants | 57 | 0

2. Primary Outcome: Number of Participants That Receive Services
Description: Based on medical record review, parent report, and 211 data, we will measure whether children are receiving intervention services, including Early Intervention or Special Education.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Telephone-based Screening | Usual Care
Number analyzed (Participants) | 77 | 75
Participants | 12 | 1

3. Secondary Outcome: Number of Participants Referred for Evaluation/Services (Early Intervention or Early Childhood Special Education)
Description: Based on medical record review, parent report, and 211 data, we measured whether any referrals were made for children with developmental or behavioral concerns, for evaluation or services.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Telephone-based Screening | Usual Care
Number analyzed (Participants) | 77 | 75
Participants | 25 | 7

4. Secondary Outcome: Primary Care Experiences: Percent of Anticipatory Guidance Topics Discussed & Percentage of Family-Centered Care Items That Participants Report as Usually or Always
Description: Based on parent interviews we will assess family experiences with primary care including receipt of recommended well-child care, using recommended anticipatory guidance and family-centered care items from the Promoting Healthy Development Survey (PHDS)
Time Frame: Baseline and 6 months
Population: Restricted to participants with parent interview at both baseline and 6-month follow-up.
Measure: Mean (Standard Deviation); unit: percentage of items
Arm/Group | Telephone-based Screening | Usual Care
Number analyzed (Participants) | 51 | 61
percentage of items
  Baseline% recommended anticipatory guidance topics | 61.0 (29.7) | 55.1 (29.1)
  Baseline% family-centered care (usually/always) | 87.2 (24.5) | 89.2 (20.5)
  6-months% recommended anticipatory guidance topics | 68.1 (26.4) | 54.6 (32.8)
  6-months% family-centered care (usually/always) | 84.9 (28.3) | 83.1 (31.1)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Telephone-based Screening | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/75
Other Adverse Events (participants affected / at risk) | 0/77 | 0/75

LIMITATIONS AND CAVEATS:
Sample of 152 children enrolled is relatively small, comes from single clinic system and was fairly homogeneous in terms of race and ethnicity, primary language, and other socio-demographic variables.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No